CLINICAL TRIAL: NCT03887273
Title: A Phase 1/2a Open-Label Study to Investigate the Safety of the Transplantation (by Injection) of Human Glial Restricted Progenitor Cells (hGRPs; Q-Cells®) Into Subjects With Transverse Myelitis (TM)
Brief Title: Study to Investigate the Safety of the Transplantation of Human Glial Restricted Progenitor Cells Into Subjects With Transverse Myelitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Q Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QTM-101
Record Dates: First submitted 2019-03-14; First posted 2019-03-22 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Transverse Myelitis
MeSH Terms: conditions — Myelitis, Transverse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Q-Cells dose level 1 (Experimental): One time surgical transplantation of Q-Cells dose level 1 unilaterally into spinal cord demyelinated lesion
  Interventions: Biological: Q-Cells
- Q-Cells dose level 2 (Experimental): One time surgical transplantation of Q-Cells dose level 2 unilaterally into spinal cord demyelinated lesion
  Interventions: Biological: Q-Cells
- Q-Cells dose level 3 (Experimental): One time surgical transplantation of Q-Cells dose level 3 unilaterally into spinal cord demyelinated lesion
  Interventions: Biological: Q-Cells

INTERVENTIONS:
Biological: Q-Cells — cellular therapeutic comprised of human cells of the glial lineage
  Other Names: glial restricted progenitor cells

SUMMARY:
This study is a non-randomized, open-label, partially blinded, sequential cohort, dose-escalation study designed to obtain preliminary data on the safety, tolerability, and early activity of Q-Cells® transplantation in subjects with Transverse Myelitis. For each of the dose levels, transplantation of Q-Cells® unilaterally into spinal cord demyelinated lesions will be evaluated. Subjects will be blinded to side of treatment.

Idiopathic Transverse Myelitis is a monophasic disorder characterized predominantly by demyelination. Patients are left with disability from damage to ascending and descending white matter tracts. Q-Cells® are comprised of glial progenitor cells.It is postulated that the Q-Cells® glial progeny (healthy astrocytes and oligodendrocytes) will integrate into the spinal cord lesion site and remyelinate demyelinated axons as well as provide trophic support for damaged axons. Therefore, Q-Cells® have the potential to repair damage that has occurred and could be clinically useful for patients with disability caused by TM.

The study is planned to enroll up to 9 subjects. Each subject will be followed for 9 months after transplantation of Q-Cells®. Each subject will receive a single time point administration of Q-Cells®: with transplantation foci targeted to posterior columns in the spinal cord (all transplantation foci below C7) on one side.

Study participation consists of Screening, Pre-operative/Treatment, and Post-treatment study periods that will generally last from 9 to 12 months in total. The study data will be assessed for safety and activity until the last subject has completed the 9-month study visit. Following completion of the 9-month follow-up period, subjects who consent will continue to be followed for safety and activity in a separate long-term follow-up protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to collect and use protected health information (PHI) in accordance with national and local subject privacy regulations.
2. Live within reasonable travel distance to center or have reliable mechanism to travel to the center.
3. Have a caregiver willing/able to assist in the transportation and care required by study participation.
4. Subject is 18 - 70 years of age (inclusive) on day of Screening Visit.
5. Subject is diagnosed with idiopathic TM within the past 120 months in accord with the Transverse Myelitis Consortium Working Group (2002).
6. Subject has a MRI with a single focus of T2 hyperintensity that is 4 to 10 cm in length if no post contrast enhancement seen, or a single focus T1 post contrast enhancing lesion of 4 to 10 cm, with its most rostral extent at or below C8 myotome/dermatome level.
7. Subject has negative NMO IgG (anti-AQP4) test at two separate time points, separated by at least 6 months.
8. Subject has brain MRI not consistent with multiple sclerosis or other autoimmune or demyelinating disease.
9. Subject is more than 12 months from TM onset.
10. Subject has ASIA A categorization.
11. Subject's neurological deficits related to TM have been stable for at least 3 months.
12. Subject is medically able to undergo the study procedures and physically able to adhere to the visit schedule at the time of study entry.
13. For women of child bearing capacity, negative pregnancy test during the Screening Period and at the Pre-Operative Visit.
14. Males and females will agree to practice effective birth control during study participation and up to one year after.

Exclusion Criteria:

1. Subject with causes of weakness, sensory loss and/or autonomic dysfunction other than TM have not been practically excluded.
2. Subject with significant cognitive impairment, clinical dementia, or major psychiatric illness including psychosis, bipolar disease, major depression, as determined by the DSM-V.
3. Subject with a diagnosis of a neurodegenerative disease (e.g., ALS, Parkinson's disease, Alzheimer's disease).
4. Subject suffering with medical conditions that impair nerve or muscle function (e.g., notable peripheral neuropathy, metabolic muscle disease) or any disease or condition that would impair the subject's neuromuscular function or impair the adequate assessment of the subject's function (e.g., severe osteoarthritis).
5. Subject with a clinically significant history of unstable cardiac, pulmonary, renal, hepatic, endocrine, hematologic, or active malignancy or infectious disease or other medically significant illness that may render them at an unacceptable risk for surgery or that may cause them to be unable to complete the scheduled duration of the trial.
6. History of spine surgery or anatomic variation incompatible with route of administration (as determined by neurosurgeon).
7. Severe spinal stenosis or cord compression causing myelopathy.
8. Abnormal flow voids on the surface of the spinal cord suggestive of arteriovenous malformation (AVM) or evidence of a vascular cause of a myelopathy (e.g., infarct of spinal artery).
9. Any evidence of CNS malignancy or clinically significant CNS lesions as defined by imaging studies of the CNS (MRI of brain and spinal cord).
10. Uncontrolled hypertension (Systolic BP>180mmHg and/or Diastolic BP >110mmHg).
11. Any history of thrombotic or embolic events.
12. Any poorly controlled medical conditions that, in the opinion of the site investigator and/or surgeon, increase risk of surgery to a medically unacceptable degree.
13. Subjects who cannot undergo MRI examination because of any contraindication to the procedure, including the presence of a pacemaker, an implanted defibrillator or certain other implanted electronic or metallic devices, or who have been or might have been exposed to metal fragments, or any reason the subject cannot undergo an MRI routinely for the duration of the trial.
14. Subject with clinically significant abnormal clinical laboratory values, as determined by the Investigator at the screening visit (Visit 1).
15. Subject who is immune compromised (by therapeutic agent or disease) or who has a condition contraindicated to treatment with immunosuppression agents (e.g., tuberculosis, latent infection) as determined by history or testing. Any subject with an ongoing infection until it has been adequately treated and it is deemed to be resolved.
16. Subject with aspartate aminotransferase (AST) or alanine aminotransferase (ALT) value >3.0 times the upper limit of normal at the screening visit (Visit 1).
17. Subject with diabetes or HgbA1c > 6.5
18. Subject with a history of alcohol or drug abuse or dependence within 1 year of screening visit (Visit 1), per DSM-V criteria.
19. Subject unlikely to comply with study requirements, as determined by Investigator.
20. Subject who has been exposed to any other experimental agent (off-label use or investigational) within 60 days of screening visit (Visit 1). Biologic agents may need additional time for washout and will be evaluated by the Sponsor on a case-by-case basis.
21. Subject with pre-existing anti-human leukocyte antigen (HLA) class I or class II antibodies directed against the Q-Cells®, as determined by panel reactive antibody (PRA) assay.
22. Allergy to study treatment or any of its constituents (e.g., chicken eggs), or allergy to any of the co-administered immunosuppressants or any of their excipients.
23. Subject with any medical condition or using concomitant medication that would contraindicate the use of tacrolimus, mycophenolate mofetil, or prednisone as determined by Investigator.
24. Subject has undergone stem cell transplantation (including T-cell or bone marrow transplants) at any time prior to study (within or outside the US).
25. Subject with evidence of deep vein thrombosis (DVT) by venous ultrasound or any previous evidence of DVT.
26. Subject has recent (1 year) or recurrent history of gastrointestinal bleeding or peptic ulcer disease or is under active treatment to prevent recurrence.
27. Subject with estimated glomerular filtration rate at screening of less than 60 mL/min/1.73m2.
28. Subjects with hereditary deficiency of hypoxanthine-guanine phosphoribosyl-transferase (HGPRT) such as Lesch-Nyhan and Kelley-Seegmiller syndrome.
29. Vaccination with live virus within 6 weeks of screening.
30. History or evidence of optic neuritis.
31. Any reason, in the judgment of the investigator, which would make the subject inappropriate for entry into this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]. | 9-months
  Safety will be measured by the number of therapy related adverse events.

SECONDARY OUTCOMES:
Scores on American Spinal Injury Association (ASIA) scale testing including motor and sensory evaluations | 9-months
  The patient's grade is based on how much sensation he or she can feel at multiple points on the body, as well as tests of motor function. Sensory grading is 0 (sensation absent), 1 (impaired sensitivity), or 2 (normal sensation) for each of light touch and pin prick sensation at each of 28 locations bilaterally: a maximum of 224 for total normal sensation. Motor function is graded from 0 (total paralysis) to 5 (normal active movement) for each of ten motor functions (e.g. knee extension; 10 total motions bilaterally) for a maximum of 100.
Quantitative muscle strength values from a hand held dynamometer (HHD) | 9-months
Pain Scores on the Visual Analog Scale (VAS) | 9-months
  VAS is a linear score where subjects rank their current pain on a scale of 0 to 10 where 0 is no pain and 10 is the worst pain imaginable.
Score on Quality of Life (QOL) Questionnaire | 9-months
  The National Institutes of Health (NIH) Patient-Reported Outcomes Measurement Information System (PROMIS) QOL questionnaire will be used to document patient reported outcomes in the following areas: Lower extremity function, Urinary/Bladder functions, Bowel functions, and Sexual functions.
Score on Ashworth Spasticity Scale | 9-months
  The Modified Ashworth Scale (MAS) will be used to measure spasticity. During the administration of the MAS the examiner passively moves the joint being tested and rates the perceived level of resistance in the muscle groups opposing the movement. The scale is single-item measures ranging from 0 to 4, where 0 indicates no increase in muscle tone and 4 indicates that the affected part is rigid in flexion or extension.
Latency and conduction velocities from tibial somatosensory evoked potentials (SSEPs) | 9-months
  Somatosensory evoked potentials (SEPs or SSEPs) are a useful, noninvasive means of assessing the somatosensory pathway functioning. Electrodes are placed on the lower extremity, the back, neck and head of a patient. A nonpainful electrical stimulus is applied to the lower extremity and the signal transduction is captured by the electrodes along the back, neck and scalp. The speed of signal transduction and amplitude of the signal is measured. Standardized values are recorded and can be monitored over time. Changes in the latency (conduction velocity) will be tracked from baseline to the 9 month outcome. Transverse Myeltitis decreases the conduction speed (an increase in latency); shorter latency (increased conduction velocity) would be an indication of recovery of function.

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No